CLINICAL TRIAL: NCT06113263
Title: The Differences Between Anterior and Posterior Decompression Surgery in Individuals with Cervical Radiculopathy and Headache - a Registry Study with 2-year Follow-up
Brief Title: Anterior and Posterior Decompression Surgery in Individuals with Cervical Radiculopathy and Headache
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jard Svensson, MSc, Linkoeping University
Other Study IDs: Dekompression_swe
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2023-11

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anterior cervical decompression surgery: Individuals underwent anterior cervical decompression surgery due to cervical radiculopathy
  Interventions: Procedure: Anterior cervical decompression surgery
- Posterior cervical decompression surgery: Individuals underwent posterior cervical decompression surgery due to cervical radiculopathy
  Interventions: Procedure: Posterior cervical foraminotomy with or without laminectomy

INTERVENTIONS:
Procedure: Anterior cervical decompression surgery — The aim of the surgery is to reduce the compression of the affected nerve. With anterior cervical decompression surgery this is achieved by removing the disc and osteophytes.
  Groups: Anterior cervical decompression surgery
Procedure: Posterior cervical foraminotomy with or without laminectomy — The aim of the surgery is to reduce the compression of the affected nerve. With posterior cervical decompression surgery more space is created for the nerve by widening the foramina where the nerve exits
  Groups: Posterior cervical decompression surgery

SUMMARY:
This is a prospective observational register-based cohort study with 2 years follow-up with data from the national Swedish Spine Register (Swespine). The aim is to study the differences between anterior and posterior decompression surgery on neck-related disability, headache, and neck- and arm pain in individuals with cervical radiculopathy and headache. Secondary, to study predictive factors for an improvement in neck-related disability, headache and neck- and arm pain after decompression srurgery. All individuals underwent either anterior or posterior decompression surgery and were operated between 2014-2021. Patient-reported data was collected preoperatively (baseline), and at 1- and 2-year follow-ups and surgeon-reported data regarding the operation were collected directly after the operation. Primary outcome is self-reported neck-related disability measured with Neck Disability Index and secondary outcomes are headache, measured with an item about headache of Neck Disability Index, and neck- and arm pain, measured with a 0 to 10-point numeric rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Underwent anterior cervical decompression surgery or posterior cervical foraminotomy with or without laminectomy for cervical radiculopathy 2014 - 2021
* Age ≥ 18 years
* Preoperatively rated 1 (I have slight headaches, which come infrequently) - 5 (I have headaches almost all the time) on an item about headache of Neck Disability Index (27)

Exclusion Criteria:

* Myelopathy
* Previous neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical radiculopathy combined with headache underwent either anterior cervical decompression surgery or posterior cervical foraminotomy
Sampling Method: Non-Probability Sample
Enrollment: 2889 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Preoperatively to 24 months follow-up
  To measure neck-specific disability; 0-100 % (0 % = no disability)

SECONDARY OUTCOMES:
Headache measured with an item of Neck Disability Index | Preoperatively to 24 months follow-up
  To measure headache; 0-5 (0 = no headache)
Numeric rating scale | Preoperatively to 24 months follow-up
  To measure neck and arm pain; 0-10 (0 = no pain)
Bakground variables | Preoperatively
  To measure gender, age, body mass index, educational level, smoker/non-smoker,
Duration of neck pain | Preoperatively
  To measure duration of neck pain; 0-4 (4 = more than 2 years) or 0-2 (2 = more than 2 years)
Duration of arm pain | Preoperatively
  To measure duration of arm pain; 0-4 (4 = more than 2 years) or 0-2 (2 = more than 2 years)
Work status | Preoperatively
  To measure the patient's work status; working (student), age retirement, sick leave, disability pension
Consumption of pain-relieving drugs | Preoperatively
  To measure the consumption of pain-relieving drugs; 0-2 (0 = no consumption)
Walking ability | Preoperatively
  To measure the walking ability; ≤ 1 km or > 1 km
Specific questions about operation data | Immediately after the operation
  To study the operation and any complications reported by the surgeon.
Self-reported other diseases that greatly limit the quality of life | Preoperatively
  To measure self-reported other diseases that greatly limit the quality of life; Yes or No (heart disease, neurological disease, cancer, others disease that limitswalking ability, other disease that causes pain)
EQ-5D-3L index | Preoperatively
  To measure health-related quality of life ; -0.594 - 1 (1 = best possible health status)

CONTACTS AND LOCATIONS:
Overall Officials: Jard Svensson, MSc, Principal Investigator — Linkoeping University

IPD SHARING:
Plan to Share IPD: No